CLINICAL TRIAL: NCT02454881
Title: Dose Response Study of Patient Controlled Analgesia (PCA) of Dexmedetomidine in Orthopaedic Spine Surgery Patients
Brief Title: Dose Response Study of Dexmedetomidine in Orthopaedic Spine Surgery Patients
Acronym: DoserespDex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T97/2015
Record Dates: First submitted 2015-05-20; First posted 2015-05-27 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Active Comparator): Oxycodone 1 mg / ml alone
  Interventions: Drug: Oxycodone
- Dexmedetomidine 2.5 (Active Comparator): Oxycodone 1 mg / mL + Dexmedetomidine 2,5 μg / mL
  Interventions: Drug: Dexmedetomidine; Drug: Oxycodone
- Dexmedetomidine 5 (Active Comparator): Oxycodone 1 mg / mL + Dexmedetomidine 5 μg / mL
  Interventions: Drug: Dexmedetomidine; Drug: Oxycodone
- Dexmedetomidine 10 (Active Comparator): Oxycodone 1 mg / mL + Dexmedetomidine 10 μg / mL
  Interventions: Drug: Dexmedetomidine; Drug: Oxycodone

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Dexdor
  Arms: Dexmedetomidine 10; Dexmedetomidine 2.5; Dexmedetomidine 5
Drug: Oxycodone
  Other Names: Oxanest

SUMMARY:
To study the multimodal protocol combining adjunct dexmedetomidine with oxycodone in intravenous patient-controlled analgesia bolus dosing and effects in patients scheduled for posterolateral lumbar spine fusion with bilateral transpedicular screw instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective posterolateral lumbar spine fusion with bilateral transpedicular screw instrumentation under general anaesthesia.
* Written informed consent from the participating subject

Exclusion Criteria:

* A previous history of intolerance to the study drug or related compounds and additives
* Concomitant drug therapy with oxycodone or buprenorphine.
* History of ischemic heart disease or conduction disturbance
* BMI > 35
* Existing significant haematological, endocrine, metabolic or gastrointestinal disease
* History of alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent
* Allergy to dexmedetomidine or oxycodone
* Blood loss exceeding 1500 ml during operation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in opioid consumption (mg) postoperatively | 24 hours
  Change from baseline opioid consumption (mg) postoperatively at 24 hours

SECONDARY OUTCOMES:
Change in numerical rating scale (NRS 0-10) | 72 hours
  Number of patients with numerical rating scale value under 3
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 72 hours
  Efficacy of dexmedetomidine as an adjuvant in postoperative analgesia with oxycodone after spinal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Teijo I Saari, MD, PhD, Principal Investigator — Dept. Anaesthesiology and Intensive Care, University Of Turku
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No